CLINICAL TRIAL: NCT04330391
Title: Implementing Weight Loss Before Total Joint Arthroplasty Using A Remote Dietitian and Mobile App: A Randomized, Control Trial
Brief Title: Weight Loss Before Total Joint Arthroplasty Using A Remote Dietitian and Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Vela Foundation (Unknown)
Responsible Party: Principal Investigator, Antonia Faustina Chen, Associate Professor of Orthopedic Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P000322
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Arthroplasties, Replacement; Weight Loss; Nutrition
Keywords: Arthroplasty; Weight loss; Health coach; dietitian
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Two group randomized control trial comparing the intervention and standard care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to the intervention or control group. The Principal Investigator and staff recording outcome measures (e.g. weighing patients) will be blinded to participant assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Individuals randomized to the usual care group will receive standard care. This may include a physical therapist and/or nutritionist referral. Brigham and Women's Hospital offers several programs for patients interested in losing weight, including the Nutrition Wellness Service (NWS) and Program for Weight Management (PWM). Insurance coverage for these programs varies by patient insurance.
- Intervention (Experimental): Intervention subjects will use the Nutrimedy mobile app and be connected at enrollment with a registered dietitian who will contact intervention participants weekly or bi-weekly via video calls and unlimited in-app text messaging for up to three months. The first week will include either one 55-minute video session or two 25-minute sessions. Weeks 2-4 will have weekly 25-minute video calls, and weeks 5-12 will have biweekly 25-minute sessions for a total of 8-9 sessions over 12 weeks. Together, participants and dietitians will come up with goals for the 12 weeks, and dietitians will check on progress toward these goals using in-app tools such as food logs and messaging between video calls. All patients will be encouraged to lose at least 20 pounds with a goal BMI<40 kg/m2 after 12 weeks. The intervention group will also receive all aspects of the usual care arm including the opportunity to have a physical therapist and/or nutritionist referral.
  Interventions: Behavioral: Remote dietitian supervised weight loss intervention and mobile app

INTERVENTIONS:
Behavioral: Remote dietitian supervised weight loss intervention and mobile app — Please see intervention arm description for more details.
  Arms: Intervention

SUMMARY:
The purpose of this trial is to assess the impact of a 12-week remote dietitian supervised dietary and physical activity weight loss intervention and mobile app for patients with morbid obesity prior to undergoing total joint arthroplasty of the hip or knee. The hypothesis is that that the intervention will result in: 1) greater weight loss than usual care, 2) a higher percentage of patients eligible to undergo surgery by having a body mass index (BMI) below the standard cutoff of 40 kg/m2, and 3) a higher percentage of patients undergoing surgery within six months of study enrollment.

DETAILED DESCRIPTION:
Recruitment: Patients of orthopaedic surgeons (e.g. Dr. Antonia Chen, Dr. Jeffrey Lange, Dr. Vivek Shah, Dr. Richard Iorio and Dr. Wolfgang Fitz) at the Brigham and Women's Hospital or Mass General Hospital orthopaedic clinics will be identified as potentially eligible for the study based on 1) 40 < body mass index (BMI) < 47 kg/m2 in the last 6 months recorded in the Partners electronic medical record, and 2) recommended unilateral total joint arthroplasty. Study flyers will be posted in MGH orthopedics clinics to remind clinicians that their patients may be eligible for the study, or patients may directly contact the research team by emailing the contact person on the flyer. For patients identified as potentially eligible while in clinic, an orthopaedic surgeon will introduce the patient to the study, and a member of the research team (research assistant or trainee) will conduct an eligibility screening (see eligibility criteria above) and obtain verbal consent either in-person or by phone. For patients identified as potentially eligible outside of clinic, a member of the research team will call the patient to introduce the study, and conduct eligibility screening and consent on the phone. Research staff may also contact these patients by email or via Patient Gateway to help coordinate a time convenient for staff to call the patient.

Interested, eligible, and consented subjects will be provisionally enrolled and each subject (both intervention and standard care participants) will be shipped a standard bathroom scale that they will keep even after the study concludes. Subjects will be asked to verify their enrollment BMI is 40 < body mass index (BMI) < 47 kg/m2. Subjects can verify weights by either a) submitting a photo to the study team of the home scale during a weigh-in that displays their body weight, or by b) recording a baseline weight at a Partners facility. For option a) subjects will submit a photo of their weight displayed on the scale to the study team either by email to a study team member's Partners email address, through the mobile app, or via RedCap. Subjects who are not able to confirm their enrollment BMI is within this range will be removed from the study. Subjects who can confirm their enrollment BMI is within this range will then be randomized to a trial arm.

Arms: Intervention participants will download the Nutrimedy telemedicine online/smartphone app and be connected at enrollment with a certified registered dietitian who will contact intervention participants weekly or bi-weekly via video calls and unlimited in-app text messaging for up to three months. The first week will include either one 55-minute video session or two 25-minute sessions. Weeks 2-4 will have weekly 25-minute video calls, and weeks 5-12 will have biweekly 25-minute sessions for a total of 8-9 sessions over 12 weeks. Together, participants and dietitians will come up with goals for the 12 weeks, and dietitians will check on progress toward these goals using in-app tools such as food logs and messaging between video calls. All patients will be encouraged to lose at least 20 pounds with a goal BMI<40 kg/m2 after 12 weeks. Intervention participants will additionally be asked if they would be interested in completing a brief 5-minute interview in-person or by phone at the end of the study (10-14 weeks after enrollment) to discuss qualitative feedback about the intervention. Responses will be transcribed verbatim during the interview for later analysis.

Individuals randomized to the usual care group will receive standard care. This may include a physical therapist and/or nutritionist referral. Brigham and Women's Hospital offers several programs for patients interested in losing weight, including the Nutrition Wellness Service (NWS) and Program for Weight Management (PWM).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age >= 18 years of age
2. BMI > 40 kg/m2 at study enrollment
3. 3. End-stage knee or hip osteoarthritis, avascular necrosis, or rheumatoid arthritis with recommended primary, unilateral total joint arthroplasty by orthopaedic surgeons at Brigham and Women's Hospital or Mass General Hospital (e.g. Dr. Antonia Chen, Dr. Jeffrey Lange, Dr. Vivek Shah, Dr. Richard Iorio and Dr. Wolfgang Fitz).
4. Subject would consider undergoing a total joint arthroplasty if eligible.
5. Owns a smartphone compatible with video calls and Nutrimedy (i.e. has access to Apple App Store or Google Play to download app) or has home internet access and a webcam for video calls.
6. All subjects must be willing to comply with the requirements of the study and provide informed consent prior to enrollment. Evidence of a signed (by the research staff obtaining verbal consent) and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study must be obtained before data collection.

Exclusion Criteria:

1. BMI>47 kg/m2 at study enrollment (BMI over 47 kg/ m2 would require inappropriate weight loss of over 3 lbs per week to reach a BMI of 40 kg/m2 after 12 weeks).
2. Subjects unable to comprehend and speak English
3. Subjects requiring a revision total joint arthroplasty
4. Subjects undergoing bilateral total joint arthroplasty
5. Subjects planning to undergo bariatric weight loss surgery in the next 6 months.
6. Subjects planning to be pregnant in the next 6 months
7. Subjects unwilling or unable to use a hand-held smartphone or personal computer with home internet access
8. Incarcerated subjects
9. Pregnant women and vulnerable individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of weight lost or gained from baseline | Final weights will be recorded at 12 weeks (10-14 weeks) after study enrollment. The baseline weight will be recorded at enrollment.
  The percentage of weight lost or gained will be determined by calculating the difference in final weight and baseline weight for each participant, divided by the baseline weight. Weights will be recorded at a Partners Healthcare facility of the patients' choice, such as at their surgeon's clinic.

SECONDARY OUTCOMES:
Percentage of patients eligible to undergo total joint arthroplasty (TJA) | This outcome will be evaluated at 3 months (10-14 weeks) after study enrollment.
  Patients are deemed eligible to undergo TJA if they have a BMI under 40 kg/m2. Weights will be recorded as described in Outcome 1.
Percentage of patients undergoing total joint arthroplasty (TJA) | This outcome will be evaluated for each subject at 6 months after study enrollment.
  Undergoing TJA will be assessed by checking participant online medical records for TJA surgery dates.
Number of completed video call sessions with dietitian | This outcome will be assessed 14 weeks after enrollment.
  Number of calls completed with a dietitian will be assessed for intervention subjects.
Change from baseline in Paving Wheel Wellness score | Baseline surveys are completed at enrollment. End-of-study surveys are assessed at 10-14 weeks after enrollment.
  Baseline and end-of-study surveys will assess behavioral, physical activity, and functional outcomes. The Paving Wheel Wellness score is calculated based on survey responses to these elements. The score ranges from 16 to 80, and a higher score indicates a better outcome.
Change from baseline in HbA1c | Baseline labs will be collected within 2 weeks of enrollment. End-of-study labs will be collected 10-14 weeks after enrollment.
  The following blood serology labs will be assessed at baseline and end-of-study: HbA1c, serum albumin, transferrin, total lymphocyte count. These labs have been recommended to assess malnutrition in orthopaedic patients.
Change from baseline in serum albumin | Baseline labs will be collected within 2 weeks of enrollment. End-of-study labs will be collected 10-14 weeks after enrollment.
  The following blood serology labs will be assessed at baseline and end-of-study: HbA1c, serum albumin, transferrin, total lymphocyte count. These labs have been recommended to assess malnutrition in orthopaedic patients.
Change from baseline in transferrin | Baseline labs will be collected within 2 weeks of enrollment. End-of-study labs will be collected 10-14 weeks after enrollment.
  The following blood serology labs will be assessed at baseline and end-of-study: HbA1c, serum albumin, transferrin, total lymphocyte count. These labs have been recommended to assess malnutrition in orthopaedic patients.
Change from baseline in total lymphocyte count | Baseline labs will be collected within 2 weeks of enrollment. End-of-study labs will be collected 10-14 weeks after enrollment.
  The following blood serology labs will be assessed at baseline and end-of-study: HbA1c, serum albumin, transferrin, total lymphocyte count. These labs have been recommended to assess malnutrition in orthopaedic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia F Chen, MD, MBA, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Statistics based on aggregated information will be published, but those statistics will not contain any Personally Identifiable Information.

REFERENCES:
- [Background] Warner DO. Surgery as a teachable moment: lost opportunities to improve public health. Arch Surg. 2009 Dec;144(12):1106-7. doi: 10.1001/archsurg.2009.205. No abstract available. PMID 20026826
- [Background] McElroy MJ, Pivec R, Issa K, Harwin SF, Mont MA. The effects of obesity and morbid obesity on outcomes in TKA. J Knee Surg. 2013 Apr;26(2):83-8. doi: 10.1055/s-0033-1341407. Epub 2013 Mar 11. PMID 23479424
- [Background] Gandler N, Simmance N, Keenan J, Choong PF, Dowsey MM. A pilot study investigating dietetic weight loss interventions and 12 month functional outcomes of patients undergoing total joint replacement. Obes Res Clin Pract. 2016 Mar-Apr;10(2):220-3. doi: 10.1016/j.orcp.2016.03.006. Epub 2016 Apr 3. PMID 27053573
- [Background] Liljensoe A, Laursen JO, Bliddal H, Soballe K, Mechlenburg I. Weight Loss Intervention Before Total Knee Replacement: A 12-Month Randomized Controlled Trial. Scand J Surg. 2021 Mar;110(1):3-12. doi: 10.1177/1457496919883812. Epub 2019 Nov 3. PMID 31679465
- [Background] Pellegrini CA, Chang RW, Dunlop DD, Conroy DE, Lee J, Van Horn L, Spring B, Cameron KA. Comparison of a Patient-Centered Weight Loss Program starting before versus after knee replacement: A pilot study. Obes Res Clin Pract. 2018 Sep-Oct;12(5):472-478. doi: 10.1016/j.orcp.2018.06.009. Epub 2018 Jul 11. PMID 30007535
- [Derived] Seward MW, Antonelli BJ, Giunta N, Iorio R, Fitz W, Lange JK, Shah VM, Chen AF. Weight loss before total joint arthroplasty using a remote dietitian and mobile app: study protocol for a multicenter randomized, controlled trial. J Orthop Surg Res. 2020 Nov 13;15(1):531. doi: 10.1186/s13018-020-02059-w. PMID 33187535